CLINICAL TRIAL: NCT04763668
Title: Assessment of the Impact of HIV Infection an Anti-retroviral Therapy (ART) on the Cardiometabolic Health of Pregnant Mothers and Their Offspring
Brief Title: Cardiometabolic Health of Children Exposed to Anti-retroviral Therapy (ART) in Utero
Acronym: ARTMOMSBABES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Walter Sisulu University (Other)
Collaborators: Nelson Mandela Academic Hospital (Unknown); Umtata General Hospital (Unknown); Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 129245
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: In Utero Drug Exposure
Keywords: ART; neonate; HIV infection; risk; cardiovascular disease; pregnant
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum from HIV infected mothers and cord blood of infants will be stored for future studies
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant HIV positive women on ART: Sub-Saharan women with singleton uncomplicated 11-14 week old pregnancies at recruitment, HIV positive and have been on ARTs for at least four months before pregnancy. Participants must not have type 2 diabetes, gestational diabetes, renal / cardiovascular diseases or any critical health condition.
  Interventions: Other: Pregnant HIV positive women on ARTs
- Pregnant HIV negative women: Sub-Saharan women with singleton uncomplicated 11-14 week old pregnancies at recruitment, HIV negative. Participants must not have type 2 diabetes, gestational diabetes, renal / cardiovascular diseases or any critical health condition.
  Interventions: Other: Pregnant HIV positive women on ARTs
- Babies born to HIV positive mothers on ARTs: All babies born to pregnant HIV positive women on ARTs who were in the first arm of the study
  Interventions: Other: Babies born to HIV positive mothers on ARTs
- Babies born to HIV negative mothers: All babies born to pregnant HIV negative women who were in the first arm of the study.
  Interventions: Other: Babies born to HIV positive mothers on ARTs

INTERVENTIONS:
Other: Pregnant HIV positive women on ARTs — Cardiovascular disease risk in pregnant HIV positive women on ARTs
  Groups: Pregnant HIV negative women; Pregnant HIV positive women on ART
Other: Babies born to HIV positive mothers on ARTs — cardiovascular disease risk in the offspring of HIV positive mothers on ARTs
  Groups: Babies born to HIV negative mothers; Babies born to HIV positive mothers on ARTs

SUMMARY:
The Human Immunodeficiency Virus (HIV) has been recently linked to increased risk for cardiovascular diseases (CVDs). The prevalence of cardiovascular diseases and its risk factor, hypertension, are very high in African communities especially in the working age group which also happens to have the bulk of young female adults in the reproductive age. Hypertension in African children is becoming a real cause for concern though its etiology remains elusive. Thanks to antiretroviral therapy (ART) use, many more infected persons live long enough to reproduce, consequently, an increasing number of children are being born to mothers who are infected with HIV. Could it be that in utero exposure of these children to HIV/ART contribute in programming them for increased risk for cardiovascular diseases thus making them more vulnerable to hypertension in childhood and adulthood? This study is aimed at exploring the possible association of in utero exposure to the HIV/ART environment and an increased risk for cardiovascular disease.

DETAILED DESCRIPTION:
I. Sample size calculation The number of participants required to show statistical significance is based on previously published studies in which vascular function was assessed in HIV patients (Agu et al., 2019). An error probability (α) of 0.05, and power (1- β) of 0.80 and an average effect size (d) of 0.5 were used to calculate the sample size (n= 64 persons). Assuming a 25% drop out rate, we will use N = (64 + (64*25)/100) = 80 mothers/group to ensure that we will have enough sample size/group to show statistical significance. Total number of participating mothers will therefore be 160 (80 cases and 80 controls) and their offspring - 160.

II. Ethical approval Ethical consent and permission to carry out the research project will be obtained from the Faculty of Health Sciences Research and Ethics Committee (HRSEC) at Walter Sisulu University (WSU). The purpose of the study will be explained to women attending the antenatal clinic in the Umtata General and Nelson Mandela Academic Hospitals, Mthatha, Eastern Cape Province. Pregnant women who will be willing to participate will be required to sign informed consent forms to participate in the study and to allow their children to participate in the study from birth.

III. Study design A prospective case control study design will be used in this study.

IV. Selection criteria Sub-Saharan women with singleton uncomplicated 11-14 week old pregnancies, be HIV positive for the case group and HIV negative for the control group. Pregnant women with type 2 diabetes, gestational diabetes, renal and cardiovascular diseases or any critical health condition will be excluded from the study

V. Experimental Plan

Work Package 1 (Pregnant women):

Three antenatal visits will be recorded for this study - These visits will be done during the first, second and third trimesters of gestation.

The following information and parameters will be assessed during each antenatal visit:

1. Baseline information: Maternal demographic, obstetric and family history of cardiovascular diseases during the first visit using a questionnaire - once off at the start of the study.
2. Anthropometric measurements: Height and weight will be determined as per recommendations of the NHANES, 2009 recommendations. BMI will be calculated using the formula weight/(height (m) x height (m)).
3. Blood pressure measurements: Office blood pressure will be measured as described by Muntner et al., (2019) in triplicates at three minutes intervals after 10 minutes of rest in the seated position. This will be followed by 24 h ambulatory blood pressure measurement for determination of day time/night time blood pressure and dipping phenotype.
4. Placental morphometry, architecture and vascularization: Uterine arteries, umbilical artery and middle cerebral artery and uterine artery mean pulsating index will be determined by ultrasound. Foetal cerebroplacental ratio will be calculated when possible.
5. Endothelial function tests: Carotid intima media thickness, pulse wave velocity and flow mediated slowing and retinal artery assessment will be measured using ultrasonography and Vicorder (Ellins, 2017). Retinal microvasculature will be studied to determine endothelial function.
6. Markers of endothelial function: Endocan, asymmetric dimethyl arginine (ADMA) and nitric oxide (NO) will be assayed using ELISA kits as per manufacturers' instructions.
7. Markers of oxidative stress: Lipid peroxidation, total antioxidant capacity and 8-hydoxyl-2-deoxyguanine (8-OHdG) will be determined using ELISA kits as per manufacturer's protocols.
8. Lipid profile indices: Total cholesterol, triglyceride, LDL cholesterol and HDL cholesterol, and oxidized LDL-cholesterol will be measured as per manufacturer's protocol.
9. Insulin Resistance: Fasting glucose, glycated haemoglobin and insulin concentrations will be determined using kits as per manufacturer's methods. The HOMA-IR formula will be used to calculate insulin resistance from fast glucose and insulin.
10. Renal function indices: glomerular filtration rate (GFR), creatinine and albumin will be determined and albumin to creatinine ratio computed.

Work Package 2 (Neonates):

During delivery, cord blood will be collected for assessment of markers of oxidative stress and endothelial function and epigenetic markers in the foetus. The following data will be collected:

1. Anthropometric measurements: The weight, length, cranial circumference of the child will be measured.
2. Blood pressure measurements: Casual blood pressure will be measured by oscillometry using disposable arm-size appropriate cuffs. Blood pressure will be measure in triplicates with five minutes intervals at least one hour after baby's meal and when baby is sleeping (Samantha et al, 2015).
3. Markers of endothelial function: Endocan, asymmetric dimethyl arginine (ADMA) and nitric oxide (NO) will be assayed using ELISA kits as per manufacturers' instructions.
4. Markers of oxidative stress: Lipid peroxidation, total antioxidant capacity and 8-hydoxyl-2-deoxyguanine (8-OHdG) will be determined using ELISA kits as per manufacturer's protocols.
5. Lipid profile indices: Total cholesterol, triglyceride, LDL cholesterol and HDL cholesterol, and oxidized LDL-cholesterol will be measured as per manufacturers protocol.
6. Insulin Resistance: cord blood glucose and insulin concentrations will be determined as per manufacturer's methods. The HOMA-IR formula will be used to calculate insulin resistance.
7. Renal function indices: glomerular filtration rate (GFR), creatinine and albumin will be determined. The Albumin to creatinine ratio will also be determined.
8. Epigenetic markers: Urine concentrations of 5-methyl-2-deoxycytidine and trimethyl histone H3K9 using Elisa kit as per manufacturer's methods.

Work Package 3 (Mothers at 3 months post-natal follow-up)

Mothers will followed up three months after delivery. During this visit no blood nor will urine samples be collected from the mothers. Urine samples will be collected from babies for measurement of CVD risk makers. The following data will be collected:

1. Anthropometric measurements: Height and weight will be determined as per recommendations of the NHANES, 2009 recommendations. BMI will be calculated using the formula weight/(height (m) x height (m)) for both mother and baby.
2. Blood pressure measurements: Office blood pressure will be measured as described by Puntner et al., (2019) in triplicates at three minutes intervals after 10 minutes of rest in the seated position. This will be followed by 24 h ambulatory blood pressure measurement for determination of day time/night time blood pressure and dipping phenotype - mother
3. Blood pressure will be measured in the baby in the supine position.
4. Endothelial function tests: Carotid intima media thickness, pulse wave velocity and flow mediated slowing and retinal artery assessment will be measured using ultrasonography and Vicorder (Ellins, 2017). Retinal microvasculature will be studied to determine endothelial function in the mother.
5. Endothelial function tests: pulse wave velocity and flow mediated slowing using the Vicorder in the baby (Ng et al, 2018).

Work Package 4 (Child):

Data will be collected from children at three, twelve and twenty four months after birth as follows:

1. Anthropometric measurements: The weight, length, cranial circumference of the child will be measured.
2. Blood pressure measurements: Casual blood pressure will be measured by oscillometry using disposable arm-size appropriate cuffs. Blood pressure will be measure in triplicates with five minutes intervals at least one hour after baby's meal and when baby is sleeping (Samantha et al, 2015).
3. Endothelial function tests: pulse wave velocity and flow mediated slowing using the Vicorder (Ng et al, 2018).
4. Markers of endothelial function: Urine samples will be collected for Endocan, asymmetric dimethyl arginine (ADMA) and nitric oxide (NO) assays using ELISA kits as per manufacturers' instructions.
5. Markers of oxidative stress: Lipid peroxidation, total antioxidant capacity and 8-hydoxyl-2-deoxyguanine (8-OHdG) will be determined in urine samples using ELISA kits as per manufacturer's protocols.
6. Renal function indices: Urine creatinine and albumin will be determined. The Albumin to creatinine ratio will also be determined.
7. Epigenetic markers: Urine concentrations of 5-methyl-2-deoxycytidine and trimethyl Histone H3K9 using elisa kit as per manufacturer's methods.
8. Endothelial function tests: pulse wave velocity and flow mediated slowing using the Vicorder (Ng et al, 2018).

ELIGIBILITY:
Inclusion Criteria:

* Cases: sub-Saharan women with singleton uncomplicated 11-14 week old pregnancies, be HIV positive and have been on ARTs for at least four months before pregnancy.

Controls: 11-14 week old pregnant HIV negative women.

Exclusion Criteria:

* Pregnant women with type 2 diabetes, gestational diabetes, renal and cardiovascular diseases or any critical health.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — The project with start with pregnant women though later on both male and female offspring will be recruited in the study.
Study Population: Sub-Saharan pregnant women of African ancestry living in South Africa
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in cardiovascular risk profile during pregnancy in pregnant HIV positive women on ARTs | March 2021 to March 2022
  Cardiovascular risk will be assessed in pregnant
Assessment of of CVD risk in offspring of HIV positive mothers on ARTs | March 2021 to March 2022
  Cardiovascular risk will be assessed in the offspring of HIV positive mothers on ART at three time point: at birth, three, twelve and twenty months after birth.

CONTACTS AND LOCATIONS:
Locations (1):
- Umtata General Hospital, Mthatha, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be shared in the form of conference presentations and published peer-reviewed articles.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From March 2021 to December 2030
Access Criteria: Permission will have to be granted by relevant stakeholders.

REFERENCES:
- [Background] Agu CE, Uchendu IK, Nsonwu AC, Okwuosa CN, Achukwu PU. Prevalence and associated risk factors of peripheral artery disease in virologically suppressed HIV-infected individuals on antiretroviral therapy in Kwara state, Nigeria: a cross sectional study. BMC Public Health. 2019 Aug 20;19(1):1143. doi: 10.1186/s12889-019-7496-4. PMID 31429736
- [Background] Ellins EA, Smith KE, Lennon LT, Papacosta O, Wannamethee SG, Whincup PH, Halcox JP. Arterial pathophysiology and comparison of two devices for pulse wave velocity assessment in elderly men: the British regional heart study. Open Heart. 2017 Dec 17;4(2):e000645. doi: 10.1136/openhrt-2017-000645. eCollection 2017. PMID 29344365
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Ng KYB, Simpson NAB, Cade JE, Greenwood DC, Mcardle HJ, Ciantar E, Alwan NA. Is infant arterial stiffness associated with maternal blood pressure in pregnancy? Findings from a UK birth cohort (Baby VIP study). PLoS One. 2018 Jul 12;13(7):e0200159. doi: 10.1371/journal.pone.0200159. eCollection 2018. PMID 30001353
- [Background] Samanta M, Mondal R, Ray S, Sabui TK, Kundu CK, Hazra A, Chatterjee K, Sarkar D. Blood pressure variation with gestational age and birth weight in Indian newborn. J Trop Pediatr. 2015 Jun;61(3):197-205. doi: 10.1093/tropej/fmv019. Epub 2015 Mar 31. PMID 25833095